CLINICAL TRIAL: NCT06302387
Title: Efficacy of Acellular Dermal Matrix Versus Tenting Technique in Peri-implant Soft Tissue Augmentation and Crestal Bone Stability: A Randomized Clinical Trial
Brief Title: Acellular Dermal Matrix Versus Tenting Technique in Peri-implant Soft Tissue Augmentation and Crestal Bone Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, German O. Gallucci, Associate Professor and Chair Department of Restorative Dentistry and Biomaterials Sciences, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BEC-LSMU(R)-27
Record Dates: First submitted 2024-02-21; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Soft Tissue Augmentation
Keywords: dental implant; phenotype; mucosal tissues; mucosal tissue augmentation; vertical soft tissue height; bone resorption; bone remodeling
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Intervention Model Description: The interventional study model for this trial is a two-arm, double-blind, randomized, prospective controlled clinical trial.
Who Masked: Participant, Care Provider
Masking Description: double-blind, where neither the patients nor the clinicians responsible for treatment know the specific treatment modality
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acellular Dermal Matrix (Experimental): This group received vertical soft tissue thickness augmentation using an acellular dermal matrix.
  Interventions: Procedure: Acellular Dermal Matrix
- Soft Tissue Expansion using Tenting Technique (Experimental): This group underwent soft tissue expansion using a tenting technique with a submerged healing abutment.
  Interventions: Procedure: Soft Tissue Expansion using Tenting Technique

INTERVENTIONS:
Procedure: Acellular Dermal Matrix — The ADM arm involved vertical soft tissue augmentation using an acellular dermal matrix. This process included the placement of a porcine dermal collagen graft (Mucoderm®, Institut Straumann AG, Switzerland) atop the dental implant site. The graft, measuring 15x20 mm, was hydrated in a 0.5% Metronidazole solution for 20 minutes before application, then trimmed and placed to extend 10 by 5 mm beyond the implant margins in both buccal and lingual directions. The primary wound closure was achieved using double mattress suturing with 6-0 Prolene (Ethicon, USA).
  Arms: Acellular Dermal Matrix
Procedure: Soft Tissue Expansion using Tenting Technique — The Tenting Technique arm involved soft tissue expansion using a submerged healing abutment to promote soft tissue growth. After implant placement, 2 mm healing abutments were set on the implants. Flaps were mobilized using vertical releasing incisions, and tension-free wound closure was achieved with horizontal mattress sutures followed by suturing the incision line with interrupted sutures for primary and submerged healing. This method aimed to create a subepithelial healing space for soft tissue expansion and augmentation.
  Arms: Soft Tissue Expansion using Tenting Technique

SUMMARY:
This study looks at two ways to make gums thicker and bones stable around dental implants for people with thin gums. It compares two methods in 40 people: one method uses a special graft, and the other uses a technique called tenting. The goal is to see which method might work better for making the gums and bones around implants healthier. The check-ups are planned when the implant is put in and again after one year. The study focuses on how these methods are done without talking about what the results are.

DETAILED DESCRIPTION:
The study's protocol entails a randomized comparison between acellular dermal matrix grafting and the tenting technique, aimed at enhancing gum thickness and bone stability around dental implants in individuals with thin gum profiles. Forty participants are systematically assigned to one of the two methods under investigation. The study is structured to evaluate the interventions' potential in improving conditions conducive to the success of dental implants, specifically targeting soft tissue thickness and crestal bone level stability. The comprehensive investigation is designed to explore effective approaches for managing patients with particular soft tissue challenges, focusing on the clinical application and procedural aspects without presenting any results or conclusions.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18-75 years old.
* Physical and psychological capacity to undergo implant therapy (ASA I or II).
* Fully healed single mandibular posterior treatment sites (premolars or molars) being edentulous for at least 3 months.
* Minimum of 6 mm width and 8 mm height native bone ridge.
* No requirement for concomitant or a history of regenerative treatments.
* Minimum of 4mm keratinized mucosa at the implant site (2 mm buccal and 2mm lingual).
* Healthy non-inflamed keratinized soft tissues with a maximum soft tissue thickness height of 2 mm measured at crestal buccal and lingual aspects.
* Periodontally healthy by fulfilling all of the following criteria: Full-mouth bleeding score (FMBS) < 20%, Full-mouth plaque score (FMPS) < 15%, Community Periodontal Index of Treatment Needs (CPITN) < 2.

Exclusion Criteria:

* Patients with a history of periodontitis.
* Poor oral hygiene after Oral Hygiene Instructions (OHI).
* Pregnant or lactating.
* Uncontrolled concomitant medical diseases, e.g., diabetes.
* Receiving or having received pharmacological treatment affecting wound healing within 3 months prior to the study-related intervention.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Crestal Bone Levels | Baseline - 1year follow up
  Assessment of changes in crestal bone level (CBL)

SECONDARY OUTCOMES:
Vertical soft tissue thickness | Measured from before implant placement to implant uncovering at 2 months
  Efficacy of vertical soft tissue thickness augmentation
PPD | Baseline - 1year follow up
  Pocket probing depth
BOP | Baseline - 1year follow up
  Bleeding on probing
PI | Baseline - 1year follow up
  Plaque Index

CONTACTS AND LOCATIONS:
Locations (1):
- VIC Clinic, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
We plan to make de-identified individual participant data (IPD) from our study on dental implant techniques available to other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Result] Linkevicius T, Linkevicius R, Alkimavicius J, Linkeviciene L, Andrijauskas P, Puisys A. Influence of titanium base, lithium disilicate restoration and vertical soft tissue thickness on bone stability around triangular-shaped implants: A prospective clinical trial. Clin Oral Implants Res. 2018 Jul;29(7):716-724. doi: 10.1111/clr.13263. Epub 2018 May 31. PMID 29855100
- [Result] Sculean A, Gruber R, Bosshardt DD. Soft tissue wound healing around teeth and dental implants. J Clin Periodontol. 2014 Apr;41 Suppl 15:S6-22. doi: 10.1111/jcpe.12206. PMID 24641001